CLINICAL TRIAL: NCT01355666
Title: Evaluate the Efficacy of a Silk-Like Fabric for the Prevention of Pressure Sores in a Long Term Care Setting
Brief Title: Silk-Like Fabric for the Prevention of Pressure Sores in a Long Term Care Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Precision Fabrics Group, Inc. (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Dr. Terry Montgomery, Precision Fabrics Group, inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DermaTherapy
Record Dates: First submitted 2011-05-13; First posted 2011-05-18 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2011-05

CONDITIONS: Pressure Ulcers
Keywords: pressure ulcers; stage 1; stage 2; stage 3; stage 4; wounds; sores; infection; bioburden; bacterial contamination; bed linen; sheets; underpad; skin assessment; microclimate; shear; friction; moisture; fabrics; long term care; nursing home; decubitus ulcer; bed ridden; anti-microbial
MeSH Terms: conditions — Pressure Ulcer; Wounds and Injuries; Infections | interventions — Absorbent Pads

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DermaTherapy® Linen group (Experimental): The DermaTherapy® Linen group uses bed sheets and underpads made with DermaTherapy® fabric.
  Interventions: Device: DermaTherapy® Linen and underpads.

INTERVENTIONS:
Device: DermaTherapy® Linen and underpads. — DermaTherapy® Linen is a 100% synthetic silk-like fabric technology designed to provide a cleaner, drier and smoother surface between the skin and support systems for a healthy micro-climate.
  Subjects in the DermaTherapy® Linen Group are compared to subjects receiving usual care - bed linen made of cotton-blend fabrics.
  Other Names: DermaTherapy®

SUMMARY:
The primary purpose of this research study is to evaluate if DermaTherapy® bedding will significantly reduce pressure ulcer incidence by decreasing maceration, friction, and shearing among residents of Nursing Homes.

DETAILED DESCRIPTION:
Additional objectives of this research study are:

* To evaluate healing of pressure ulcers already present or pressure ulcers that develop during the study.
* To evaluate the effectiveness of DermaTherapy® bedding and alternative diapers to reduce the potential for bacterial contamination associated with patients' bed linens, underpads, gowns and pajamas, and thereby help reduce the incidence of facility-acquired infections.

Study nurses will assess the skin of the subjects once or twice a week for the presence of pressure ulcers and measure the size of the pressure ulcers if they are present. Study nurses will also obtain bacterial culture swabs of the bedding weekly for the first eight weeks of the study from five participants in each group.

ELIGIBILITY:
Inclusion Criteria:

* Residents admitted for long term care.
* Residents admitted for Hospice Care with an expected length of stay greater than one week.
* Residents with an expected length of stay equal to or greater than 90 days.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-05 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Prevention and reduction in the incidence of pressure ulcers | Weekly assessments for 1 year
  The primary purpose of this research study is to evaluate if DermaTherapy® bedding will significantly reduce pressure ulcer incidence by decreasing maceration, friction, and shearing among residents of Nursing Homes.

SECONDARY OUTCOMES:
Reduction of bacterial contamination | Weekly for 8 weeks
  To evaluate the effectiveness of DermaTherapy® bedding to reduce the potential for bacterial contamination associated with patients' bed linens and thereby help reduce the incidence of facility-acquired infections.

CONTACTS AND LOCATIONS:
Overall Officials: Jack I Twersky, MD, Principal Investigator — Durham VA Medical Center, Duke University Medical Center; Kenneth E Schmader, MD, Principal Investigator — Durham VA medical Center, Duke University Medical Center
Locations (1):
- Durham VA Medical Center, Durham, North Carolina, United States